CLINICAL TRIAL: NCT03521414
Title: The Effect of Glasgow Coma Scales on General Anesthesia in Neurosurgery Patients
Brief Title: Glasgow Coma Scales and General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Sevtap Hekimoglu Sahin, Director, clinical research, Trakya University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: TÜTF-GOKAEK 2013/127
Record Dates: First submitted 2018-04-24; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Anesthesia Awareness
Keywords: Bispectral index; Glasgow Coma Scale; intracranial pathology
MeSH Terms: conditions — Intraoperative Awareness | interventions — Sevoflurane

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I=13-15 mildly injured (Active Comparator): Patients were divided into 3 groups according to the Glasgow Coma Scores calculated before surgery. use of anesthetic agent were recorded during bispectral index (BIS) monitoring and anesthesia application. we used sevoflurane drug intraoperative.
  Group I (n=15)=13-15 mildly injured
  Interventions: Device: Bispectral index (BIS) monitoring; Drug: Sevoflurane
- Group 2 =9-12 moderately damaged (Active Comparator): Patients were divided into 3 groups according to the Glasgow Coma Scores calculated before surgery.use of anesthetic agent were recorded during bispectral index (BIS) monitoring and anesthesia application. we used sevoflurane drug intraoperative.
  Group 2 (n=15)=9-12 moderately damaged
  Interventions: Device: Bispectral index (BIS) monitoring; Drug: Sevoflurane
- Group 3=3-8 severely damaged. (Active Comparator): Patients were divided into 3 groups according to the Glasgow Coma Scores calculated before surgery. use of anesthetic agent were recorded during bispectral index (BIS) monitoring and anesthesia application. we used sevoflurane drug intraoperative.
  Group 3 (n=15)=3-8 severely damaged.
  Interventions: Device: Bispectral index (BIS) monitoring; Drug: Sevoflurane

INTERVENTIONS:
Device: Bispectral index (BIS) monitoring — When the patients were taken to the operation table, they were monitored with the BIS. we used sevoflurane drug
Drug: Sevoflurane — we used sevoflurane drug at inoperative

SUMMARY:
The study evaluates the general anesthesia management with BIS monitorization in terms of hemodynamic stability, drug concentrations and drug consumption in patients who underwent surgery due to intracranial pathology and who were divided in three different GCS groups.

DETAILED DESCRIPTION:
BIS monitoring is mostly used for anesthesia depth and sedation level follow-up, however it can also be used for monitoring consciousness after resuscitation of cases with acute brain injury and cardiac arrest. It is not always possible to monitor and objectively measure the changes in the level of consciousness in clinical practice. Therefore, device-based methods have been introduced in monitoring the state of consciousness. Bispectral index (BIS) monitoring may be preferred in follow up of the state of consciousness in critical patients such as those with acute brain injury, in terms of ease of use, ability to obtain numerical results and continuous monitoring. BIS monitoring is mostly used for follow up of anesthesia depth and sedation level, while it can also be applied for monitoring state of consciousness following resuscitation in cases with acute brain injury and cardiac arrest.In this study, we aimed to investigate general anesthesia management performed by bispectral index monitoring in patients who underwent surgery due to intracranial pathology and with different Glasgow Coma Scales.

ELIGIBILITY:
Inclusion Criteria:

* 18 and 65 years
* ASA II-III
* intracranial surgery

Exclusion Criteria:

* Patients with additional disease (electrolyte impairment, uremia, etc.),
* liver and renal failure affecting consciousness level other than intracranial pathology

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-07-03 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-11-05 (Actual)

PRIMARY OUTCOMES:
BIS, Consumption of the inhalation agents | 200 minutes
  Preoperative, intraoperative and postoperative BIS values were recorded. The total
  amount of opioid consumed was recorded from the infusion pump.

IPD SHARING:
Plan to Share IPD: No